CLINICAL TRIAL: NCT04104308
Title: Association of Egg and Dietary Cholesterol Consumption With Mortality and Metabolic Syndrome
Brief Title: Association of Egg and Dietary Cholesterol Consumption With Mortality and Diseases
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Jingjing Jiao, Associate Professor, Zhejiang University
Other Study IDs: Cohort_egg_mortality
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Mets; Death
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The blood samples were collected in 2009 for the first time
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess the associations between egg and dietary cholesterol consumption with mortality and metabolic syndrome (MetS).

DETAILED DESCRIPTION:
Substitution models, sensitivity analyses, subgroup analyses and multiple linear regression analyses will be conducted to specifically estimate the hazard ratios and 95% confidence intervals of mortality and MetS associated with egg and cholesterol consumption.

ELIGIBILITY:
Inclusion Criteria:

* participants aged ≥20 y

Exclusion Criteria:

* missing creatinine, age, cannot be linked to socio-demographic data; aged less than 20; without complete dietary data .

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The CHNS is a nationwide cohort survey in China, which was established as a joint project of the University of North Carolina at Chapel and the China Center for Disease Control and Prevention (CCDC).This national-wide survey adopted a novel measure from multiple dimensions, which helped to understand how the long-term social and economic changes affected nutrition and health-related outcomes of Chinese. Until now, 10 rounds of survey (1989, 1991, 1993, 1997, 2000, 2004, 2006, 2009, 2011 and 2015) have been conducted.
Sampling Method: Probability Sample
Enrollment: 33453 (Actual)
Dates: Start 1991-01-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
mortality | participants were followed up from 1991 to 2015
  mortality

SECONDARY OUTCOMES:
metabolic syndrome | The blood samples were collected in 2009 for the first time.
  MetS was defined according to the updated National Cholesterol Education Program Adult Treatment Panel III (NCEP: ATP III) criteria for Asian-Americans.

REFERENCES:
- [Derived] Wu F, Zhuang P, Zhan C, Shen X, Jiao J, Zhang Y. Egg and Dietary Cholesterol Consumption and the Prevalence of Metabolic Syndrome: Findings from a Population-Based Nationwide Cohort. J Acad Nutr Diet. 2022 Apr;122(4):758-770.e5. doi: 10.1016/j.jand.2021.09.010. Epub 2021 Oct 11. PMID 34506988
- [Derived] Zhuang P, Jiao J, Wu F, Mao L, Zhang Y. Egg and egg-sourced cholesterol consumption in relation to mortality: Findings from population-based nationwide cohort. Clin Nutr. 2020 Nov;39(11):3520-3527. doi: 10.1016/j.clnu.2020.03.019. Epub 2020 Mar 28. PMID 32307193